CLINICAL TRIAL: NCT01841437
Title: Glaukos® iStent® Trabecular Micro-Bypass Stent System In Conjunction With Cataract Surgery Postmarket Registry
Status: Completed | Type: Observational
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: GTS100-PAR
Record Dates: First submitted 2013-04-24; First posted 2013-04-26 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-08

CONDITIONS: Primary Open-angle Glaucoma
Keywords: Primary open-angle glaucoma (POAG); Trabecular meshwork; iStent
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- iStent
  Interventions: Device: iStent

INTERVENTIONS:
Device: iStent

SUMMARY:
The purpose of this study is to observe the safety of the Glaukos® iStent® Trabecular Micro-Bypass Stent Model GTS100 in conjunction with cataract surgery in subjects with mild to moderate open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive subjects in whom implantation of the iStent is attempted

Exclusion Criteria:

* Please refer to approved indications in Directions for Use

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive subjects in whom implantation of the iStent is attempted at selected clinical sites
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2013-09; Primary Completion 2016-02-16 (Actual); Study Completion 2016-06-21 (Actual)

PRIMARY OUTCOMES:
Rate of sight-threatening adverse events | 36 months

SECONDARY OUTCOMES:
Other ocular adverse events | 36 months

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Chico, California
  - Huntington Beach, California
  - Napa, California
  - Santa Maria, California
  - Ventura, California
  - Parker, Colorado
  - Portland, Maine
  - Quincy, Massachusetts
  - Bloomington, Minnesota
  - Westwood, New Jersey
  - Durham, North Carolina
  - Fayetteville, North Carolina
  - Southern Pines, North Carolina
  - Brecksville, Ohio
  - Youngstown, Ohio
  - Ladson, South Carolina
  - Sioux Falls, South Dakota
  - Appleton, Wisconsin